CLINICAL TRIAL: NCT01944046
Title: Phase II Study of Oxytocin in Autism to Improve Reciprocal Social Behaviors
Brief Title: Study of Oxytocin in Autism to Improve Reciprocal Social Behaviors
Acronym: SOARS-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Linmarie Sikich (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Linmarie Sikich, Associate professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00063950; 1U01HD073984 (NIH); 13-0593 (Other: UNC)
Record Dates: First submitted 2013-06-13; First posted 2013-09-17 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Autism Spectrum Disorders
Keywords: autism, ASD, autistic, Asperger's, PDD-NOS, oxytocin
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, placebo-controlled clinical trial for 24 weeks. Followed by 24 week open label treatment period in which ALL participants receive Oxytocin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DB Placebo Nasal Spray (Placebo Comparator): Placebo treatment during weeks 0-24 double blind phase
  Interventions: Drug: Double blind phase Placebo Nasal Spray
- DB Oxytocin Nasal Spray (Active Comparator): DB Oxytocin- quadruply masked treatment with intranasal oxytocin during weeks 0-24 of study during double blind phase of study
  Interventions: Drug: double Blind Oxytocin Nasal Spray
- open label intranasal oxytocin (Active Comparator): non masked treatment with intranasal oxytocin from weeks 24-48 in those participants who completed first 24 weeks of double blind treatment
  Interventions: Drug: Open Label intranasal oxytocin

INTERVENTIONS:
Drug: Double blind phase Placebo Nasal Spray — This nasal spray will contain all of the ingredients that are in the active oxytocin spray in the same quantities, except oxytocin will NOT be added to the solution. It will be packaged using the same container system as the active oxytocin nasal spray. Each bottle's label will have its own unique nonsequential randomly assigned number and not a lot number to facilitate masking. Dose titration will occur using exactly the same criteria and procedures as for active study drug.
  Other Names: DB Placebo (PL)
  Arms: DB Placebo Nasal Spray
Drug: double Blind Oxytocin Nasal Spray — Each insufflation will deliver 8 IU or 24 IU of oxytocin. A maximum of 3 insufflations at a time will be required. Dosing will be flexible between 8 IU/day and 80 IU/day, typically in two divided doses delivered in the morning and in the afternoon. Doses will typically increase by 8 IU twice daily (BID) at week 2 and weeks 4 and 8 until achieving the target dose of 24 IU BID at week 8. Subsequently doses may be increased in 8 IU BID increments ONLY at each visit until a maximum dose of 40 IU BID is achieved.Each bottle's label will have its own unique nonsequential randomly assigned number and not a lot number to facilitate masking. During the open label phase after approximately March 2019 the study used only the 24 IU /0.10 ml formulation and the maximum dose was 72 IU per day.
  Other Names: DB Intranasal Oxytocin (OT)
  Arms: DB Oxytocin Nasal Spray
Drug: Open Label intranasal oxytocin — All participants who completed the 24 week double blind phase were eligible to join a 24 week open label phase in which all participants received intranasal oxytocin
  Other Names: open label treatment
  Arms: open label intranasal oxytocin

SUMMARY:
The purpose of this research study is to learn about the effects of supplemental intranasal oxytocin as a treatment for improving social difficulties in children and adolescents with autism. This study will also provide additional information about the safety and tolerability of intranasal oxytocin. Investigators expect oxytocin will increase social motivation, improving daily living skills and quality of life.

DETAILED DESCRIPTION:
There is a tremendous unmet need for accessible treatments that address core symptoms of ASD and are safe for sustained use. The Study of Oxytocin in ASD to improve Reciprocal Social Behaviors or (SOARS-B) will test a very promising potential treatment-intranasal oxytocin-for ASD's fundamental social communication deficits in a large, group of verbal and nonverbal children. SOARS-B will also provide information about the regulation of DNA methylation and transcription of the oxytocin receptor gene (OXTR), as well as other genes relevant to oxytocin's CNS activity, as a function of time and in response to oxytocin treatment. These data will fill a key gap in our understanding of oxytocin's role in ASD and its ability to alter epigenetic modifications of the OXTR.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 3 years 0 months and 17 years 11 months at the time of randomization
* Be diagnosed by clinician experienced in assessment of ASD with autistic disorder, Asperger's syndrome, or PDD-NOS using DSM-V-TR criteria
* Must have clinical diagnosis of ASD confirmed using the Autism Diagnostic Observation Scale (ADOS, Lord et al., 2001)
* Must have clinical diagnosis of ASD confirmed using the Autism Diagnostic Interview-Revised (ADI-R, Rutter, 2003). ASD criteria proposed by Risi (2006). Specifically, subject must be within 1 point of autism criteria on both social and communication domains of the ADI or meet autism criteria in one of these ADI domains and come within 2 points of autism criteria in the other
* Have a guardian who is able to provide informed consent
* If cognitively able, subject must be able to provide informed assent/consent

Exclusion Criteria:

* Have a known diagnosis of Rett Syndrome or Childhood Disintegrative Disorder, or have marked sensory impairment such as deafness or blindness
* Have active cardiovascular disease or renal disease that is not controlled by medication
* Subjects who are pregnant, lactating, or who refuse to practice contraception if sexually active
* Subjects who have had changes in allied health therapies, behavioral or educational interventions within the two months prior to randomization other than those associated with school holidays
* Subjects who have had changes in psychiatric medications within 4 weeks of randomization
* Subjects who have had previous chronic treatment with oxytocin
* Subjects who have caretakers who are unable to speak English, be consistently present at visits to report on symptoms, or are otherwise judged as unable to comply with the protocol by the data collection site team
* Subjects with active seizures within the 6 months preceding screening or baseline -added part way through study in response to subject death.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Lurie Center for Autism, Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - Center for Autism and the Developing Brain, White Plains, New York
  - Duke Center for Autism and Brain Development, Durham, North Carolina
  - Duke University , Genetics Center, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Seattle Children's Hospital Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Most data will be available on NDAR, but will not be identifiable.

REFERENCES:
- [Background] Spanos M, Chandrasekhar T, Kim SJ, Hamer RM, King BH, McDougle CJ, Sanders KB, Gregory SG, Kolevzon A, Veenstra-VanderWeele J, Sikich L. Rationale, design, and methods of the Autism Centers of Excellence (ACE) network Study of Oxytocin in Autism to improve Reciprocal Social Behaviors (SOARS-B). Contemp Clin Trials. 2020 Nov;98:106103. doi: 10.1016/j.cct.2020.106103. Epub 2020 Aug 8. PMID 32777383
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Sikich L, Kolevzon A, King BH, McDougle CJ, Sanders KB, Kim SJ, Spanos M, Chandrasekhar T, Trelles MDP, Rockhill CM, Palumbo ML, Witters Cundiff A, Montgomery A, Siper P, Minjarez M, Nowinski LA, Marler S, Shuffrey LC, Alderman C, Weissman J, Zappone B, Mullett JE, Crosson H, Hong N, Siecinski SK, Giamberardino SN, Luo S, She L, Bhapkar M, Dean R, Scheer A, Johnson JL, Gregory SG, Veenstra-VanderWeele J. Intranasal Oxytocin in Children and Adolescents with Autism Spectrum Disorder. N Engl J Med. 2021 Oct 14;385(16):1462-1473. doi: 10.1056/NEJMoa2103583. PMID 34644471

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxytocin Nasal Spray: Oxytocin
  Oxytocin Nasal Spray: Each insufflation will deliver 8 IU or 24 IU of oxytocin. A maximum of 3 insufflations at a time will be required. Dosing will be flexible between 8 IU/day and 80 IU/day, typically in two divided doses delivered in the morning and in the afternoon. Doses will typically increase by 8 IU twice daily (BID) at week 2 and weeks 4 and 8 until achieving the target dose of 24 IU BID at week 8. Subsequently doses may be increased in 8 IU BID increments ONLY at each visit until a maximum dose of 40 IU BID is achieved.Each bottle's label will have its own unique nonsequential randomly assigned number and not a lot number to facilitate masking. During the open label phase after approximately March 2019 the study used only the 24 IU /0.10 ml formulation and the maximum dose was 72 IU per day.
- Placebo Nasal Spray: Placebo
  Placebo Nasal Spray: This nasal spray will contain all of the ingredients that are in the active oxytocin spray in the same quantities, except there will be no oxytocin added to the solution. It will be packaged using the same container system as the active oxytocin nasal spray. Each bottle's label will have its own unique nonsequential randomly assigned number and not a lot number to facilitate masking. Dose titration will occur using exactly the same criteria and procedures as for active study drug.
Period: Randomized to DB
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Started | 146 | 144
Completed | 125 | 125
Not Completed | 21 | 19
Not completed — Adverse Event | 5 | 2
Not completed — Clinical Worsening | 3 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 1 | 2
Not completed — Did not have baseline ABC-SW | 2 | 0
Not completed — Did not have a postbaseline ABC SW | 5 | 6
Period: Open Label Eligible and Consented
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Started (1 from each treatment group declined to consent for openlabel) | 124 | 124
Completed | 110 | 116
Not Completed | 14 | 8
Not completed — Lost to Follow-up | 3 | 5
Not completed — Adverse Event | 6 | 1
Not completed — Clinical Worsening | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Double-Blind Full Analysis Set (FAS). The DB FAS was defined as having both baseline and at least one post-baseline ABC-SW assessment. The DB-FAS excludes 7 participants randomized to oxytocin (2 with no baseline ABC-SW and 5 with no post-baseline ABC-SW) and 6 participants assigned to placebo who had no post-baseline ABC-SW.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 139 | 138 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (4.06) | 10.4 (3.99) | 10.4 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 122 | 120 | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 28
  Not Hispanic or Latino | 126 | 123 | 249
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 14 | 23
  White | 104 | 100 | 204
  More than one race | 14 | 9 | 23
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139 | 138 | 277
Aberrant Behavior Checklist Social Withdrawal Subscale Score (ABC-SW) abc-SW (mean [Mean (Standard Deviation); unit: units on a scale] — the Aberrant Behavior Scale Social withdrawal score assesses reciprocal social behaviors. It is composed of 13 questions from the Aberrant Behavior Scale Lethargy subscale that consists of 16 questions. The ABC-SW does not include the 3 questions (i.e. 3,32,53) of the Lethargy subscale that refer to sedentary behaviors. Score for each item ranges from 0 (not at all a problem) to 3 (a serious problem). Items are summed to give a minimal score of 0 and a maximal score of 39. Lower Scores are better
  units on a scale | 11.0 (6.9) | 11.6 (7.8) | 11.3 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Aberrant Behavior Checklist-Modified Social Withdrawal Subscale ABC-mSW, a Measure of Social Reciprocity
Description: The primary outcome is Change in Aberrant Behavior Checklist-Modified Social Withdrawal subscale- a measure of reciprocal social behaviors. ABC-mSW is a modification of the ABC-Lethargy subscale. The ABC-mSW consists of the sum of questions 5,12,16, 20, 23, 26, 30, 37, 40, 42, 43, 55, and 58. In contrast to the ABC-Lethargy subscale it eliminates question 3 (listless, sluggish, inactive), question 32 (sits or stands in one position for a long time), and question 53 (inactive, never moves spontaneously). Thirteen individual items are scored 0-3, therefore the range is 0-39. Higher score indicates lower social reciprocity. Repeated measures were obtained at baseline, weeks 4, 8, 12, 16, 20, 24.
Time Frame: Least Mean Squares Double-blind phase: change from baseline to week 24
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale
  Double-blind baseline to w4 | 8.81 (0.39) | 8.68 (0.39)
  Double-blind baseline to w8 | 8.97 (0.45) | 8.68 (0.45)
  Double-blind baseline-w12 | 7.48 (0.43) | 8.13 (0.43)
  DB w0- w16 | 7.99 (0.46) | 8.04 (0.46)
  DB w0- w20 | 7.81 (0.05) | 7.75 (0.45)
  DB w0-w24 | 7.75 (0.46) | 8.05 (0.46)
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Superiority; p = 0.503, Mixed Models Analysis — not adjusted primary outcome; adjusted for baseline, age category, functionality category

2. Primary Outcome: Change in Aberrant Behavior Checklist-Modified Social Withdrawal Subscale ABC-mSW, a Measure of Social Reciprocity
Description: The ABC-mSW is described above and involves 13 items reflecting lack of reciprocal interaction. Each item is scored from 0 (never shows behavior) to 3 (behavior is a major problem). The range is 0-39. Higher scores indicate worse reciprocal social functioning.
Time Frame: Least mean squares for Open Label: Change between weeks 24-48
Population: Open Label phase participants in OLE FAS excluding 2 participants without usable ABC-sws (either w24 or at least one pw24 ABC-sw.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 125 | 122
score on a scale
  Open Label week 24 | 7.83 [7.11 to 8.55] | 7.81 [7.09 to 8.52]
  Open Label week 48 | 6.99 [6.10 to 7.89] | 6.78 [5.89 to 7.67]
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Superiority; p = 0.61, Mixed Models Analysis — not adjusted primary outcome, p threshold 0.05; adjustment for value at week 24,

3. Secondary Outcome: Change in Sociability Factor (SF)
Description: The Sociability Factor (SF) is a summed measure of the13 items of the ABC-SW and the 18 items of the Pervasive Development Disorders Behavior Inventory-Screening Version (PDDBI-SV).The PDDBI-SV assesses both adaptive social behaviors and social problems typical of ASD. The adaptive behaviors are reverse scored so that all the analyzed scores range from 0-performing in a neurotypical fashion to 3 typically performs in a way associated with ASD. the total # of items on this summed measure is 31 with a range from 0 to 93. More impaired social functioning indicated by higher scores. This measure was changed to a secondary outcome in the final statistical analysis plan.
Time Frame: Double-blind phase: change in least means squares between week 0 & 24.
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale
  DB w0 | 35.8 (1.24) | 36.1 (1.28)
  DB w0-w4 | -5.57 (0.69) | -5.81 (0.69)
  DB w0-w8 | -5.99 (0.66) | -6.30 (0.66)
  DB w0-w12 | -6.40 (0.66) | -6.79 (0.66)
  DB w0-w16 | -6.82 (0.70) | -7.28 (0.71)
  DB w0-w20 | -7.24 (0.88) | -7.77 (0.88)
  DB w0-w24 | -7.66 (0.78) | -8.27 (0.88)

4. Secondary Outcome: Change in Social Responsiveness Scale-2 (SRS-2) Social Motivation Subscale Score
Description: The SRS-Social Motivation subscale was developed to provide a quantitative measure of social impairments typically observed in ASD in children 3-18 years. Reported as T-score with a range of 38-90 for both boys and girls. Higher score indicates more severe clinical condition. Lower value in change indicates more improvement.
Time Frame: Double-blind phase: baseline, weeks 12, 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
T-score
  Double-blind baseline to week 12 | -4.58 (0.68) | -5.72 (0.69)
  Double-blind baseline to week 24 | -4.49 (0.70) | -5.42 (0.70)

5. Secondary Outcome: Change in Stanford Binet-5th Edition (SB-5) IQ Score
Description: Cognitive skills will be assessed using the Stanford Binet-5th Edition (SB-5) (Roid). Acceptable IQ range is 47-153, with higher score being better. Higher change scores indicate more improvement.
Time Frame: Double-blind phase: baseline to week 24
Population: Participants with scores collected at baseline and week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 94 | 98
score on a scale | 0.40 (11.64) | 1.0 (10.84)

6. Other Pre Specified Outcome: Social Responsiveness Scale-2 (SRS-2) Social Motivation Subscale Score
Description: as for outcome 4
Time Frame: Open Label: weeks 24, 48
Population: Open Label phase participants
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 127 | 122
T-score
  Open Label week 24 | 88.5 (1.37) | 86.6 (1.37)
  Open Label week 48 | 87.9 (1.83) | 83.0 (1.81)

7. Other Pre Specified Outcome: Change in Vineland II Adaptive Behavior Scales (VABS-II) Daily Living Domain Score
Description: Functional skills will be assessed using the VABS-II Daily Living Domain Score. Uses standard score with a mean of 100 and SD of 15 with a range of 20-160. Higher score is better. Higher value in change indicates more improvement.
Time Frame: Double-blind phase: baseline, week 24; Open Label: week 48
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale
  Double-blind baseline to week 24 | 2.50 (1.10) | 1.24 (1.14)
  Open Label week 24 to week 48: number analyzed (Participants) | 127 | 122
  Open Label week 24 to week 48 | 1.76 (1.19) | 0.62 (0.11)

8. Other Pre Specified Outcome: Caregiver Strain Questionnaire (CSQ) Subjective Internalizing Subscale Mean Score
Description: Caregiver questionnaire that assesses the impact of caring for the proband on caregiver and family. Each item on the subjective internalizing CSQ subscale is rated from 1 to 5. Then all items within the subscale are summed and the mean is determined based on the number of items in the subscale. Higher score indicates more caregiver strain. Lower value in change indicates more improvement.
Time Frame: Open Label: weeks 24, 48
Population: Full Analysis Set participants who entered double blind and have values at week 24 AND 48
Measure: Mean (Standard Deviation); unit: mean score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 110 | 119
mean score on a scale
  Open Label week 24 | 2.96 (0.99) | 2.85 (1.00)
  Open Label week 48 | 2.97 (0.99) | 2.85 (0.97)

9. Other Pre Specified Outcome: Change in Vineland II Adaptive Behavior Scales (VABS-II) Communication Domain Score
Description: Functional skills will be assessed using the VABS-II Communication Domain Score. Uses standard score with a mean of 100 and SD of 15 with a range of 20-160. Higher score is better. Higher value in change indicates more improvement.
Time Frame: Double-blind phase: baseline, week 24; Open Label: week 48
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale
  Double-blind baseline to week 24 | 3.88 (0.89) | 2.27 (0.90)
  Open Label week 24 to week 48: number analyzed (Participants) | 127 | 122
  Open Label week 24 to week 48 | 4.06 (1.35) | 5.98 (1.41)

10. Other Pre Specified Outcome: Change in Caregiver Strain Questionnaire (CSQ) Subjective Internalizing Subscale Score
Description: Caregiver questionnaire that assesses the impact of caring for the proband on caregiver and family. CSQ subscale scores are ranged from 1 to 5. with each item of the subscale having the same range, the sum of the items within the subscale are summed, and the mean score is determined (I.e. a single # between 1 and 5) and reported. Higher scores indicate more caregiver strain. Lower value in change indicates more improvement.
Time Frame: Double-blind phase: baseline, week 24
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale | -0.16 (0.07) | -0.29 (0.07)

11. Other Pre Specified Outcome: Change in Vineland II Adaptive Behavior Scales (VABS-II) Socialization Domain Score
Description: Functional skills will be assessed using the VABS-II Socialization Domain Score. Uses standard score with a mean of 100 and SD of 15 with a range of 20-160. Higher score is better. Higher value in change indicates more improvement.
Time Frame: Double-blind phase: baseline, week 24; Open Label: week 48
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale
  Double-blind baseline to week 24 | 4.45 (1.27) | 4.87 (1.25)
  Open Label week 24 to week 48: number analyzed (Participants) | 127 | 122
  Open Label week 24 to week 48 | 1.59 (1.11) | 0.54 (1.10)

12. Other Pre Specified Outcome: Change in Caregiver Strain Questionnaire (CSQ) Objective Subscale Score
Description: Caregiver questionnaire that assesses the impact of caring for the proband on caregiver and family. CSQ subscale scores are ranged from 1 to 5. Higher score indicates more caregiver strain. Lower value in change indicates more improvement. The analysis directions for the instrument that are used in these analyses are the mean of all the responses in the scale or subscale.
Time Frame: Double-blind phase: baseline, week 24; Open Label: week 48
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale
  Double-blind baseline to week 24 | -0.16 (0.06) | -0.22 (0.06)
  Open Label week 24 to week 48: number analyzed (Participants) | 110 | 119
  Open Label week 24 to week 48 | 0.13 (0.06) | 0.44 (0.08)

13. Other Pre Specified Outcome: Change in Caregiver Strain Questionnaire (CSQ) Subjective Externalizing Subscale Score
Description: Caregiver questionnaire that assesses the impact of caring for the proband on caregiver and family. CSQ subscale scores are ranged from 1 to 5. Higher score indicates more caregiver strain. Lower value in change indicates more improvement.
Time Frame: Double-blind phase: baseline, week 24; Open Label: week 48
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale
  Double-blind baseline to week 24 | -0.08 (0.04) | -0.04 (0.04)
  Open Label week 24 to week 48: number analyzed (Participants) | 110 | 119
  Open Label week 24 to week 48 | 0.01 (0.07) | 0 (0.08)

14. Other Pre Specified Outcome: Change in Vineland II Adaptive Behavior Scales (VABS-II) Composite Score
Description: Functional skills including communication will be assessed using the VABS-II Adaptive Behavior Composite Score. Uses standard score with a mean of 100 and SD of 15 with a range of 20-160. Higher score is better. Higher value in change indicates more improvement.
Time Frame: Double-blind phase: baseline, week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 139 | 138
score on a scale | 2.61 (1.26) | 1.50 (1.27)

15. Other Pre Specified Outcome: Change in Clinical Global Impressions -Improvement Score (CGI-I)
Description: The Clinical Global Impressions - Improvement score and Severity score, which is routinely used in pharmacologic clinical trials, will capture the study physician's global impression of response. scores of 1 and 2 are considered as a percentage of total subjects in arm
Time Frame: Double blind phase: change from Baseline to week 12, and week 24. Open label phase change from week 24 to week 48
Population: full analysis set
Measure: Number; unit: percentage of participants in arm
Groups:
- Placebo Nasal Spray: Placebo
  Placebo Nasal Spray: This nasal spray will contain all of the ingredients that are in the active oxytocin spray in the same quantities, except oxytocin will NOT be added to the solution. It will be packaged using the same container system as the active oxytocin nasal spray. Each bottle's label will have its own unique nonsequential randomly assigned number and not a lot number to facilitate masking. Dose titration will occur using exactly the same criteria and procedures as for active study drug.
Arm/Group | Placebo Nasal Spray | Oxytocin Nasal Spray
Number analyzed (Participants) | 138 | 139
percentage of participants in arm | 64 | 53

16. Other Pre Specified Outcome: Reading Mind in the Eyes Test is an Objective Measures of the Extent to Which Verbal Participants With Rudimentary Knowledge of Emotion Names Are Able to Correctly Identify the Emotion Shown in a Black and White Picture of the Eyes and Nose of an Actor.
Description: This computerized task consists of a series of pictures of eyes in which the participant needs to determine which emotion the eyes are expressing from 4 emotions listed along with the picture. The outcome is the % of pictures with correct emotion identified. The range is 0 to 100%. The larger percent identified correctly indicates better ability to perceive emotions. An increase or positive change indicates better ability to identify emotions since baseline.
Time Frame: Double blind phase: change from Baseline and week 24. Note: only those who demonstrated understanding of these concepts were included in sample.
Population: only subjects who could define feelings from fluently verbal subgroup
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 69 | 64
percentage of correct responses
  DB w0 | 51.1 (18.76) | 48.2 (18.61)
  DB w24 | 54.9 (14.02) | 49.92 (13.84)

ADVERSE EVENTS:
Time Frame: Through post-treatment follow-up, approximately 55 weeks.
Description: Adverse events collected on Safety Population (subjects who started each phase).
Groups:
- Oxytocin Nasal Spray: Double-blind Phase; Oxytocin Nasal Spray: Open Label Phase: Oxytocin
  Oxytocin Nasal Spray: Each insufflation will deliver 8 IU or 24 IU of oxytocin. A maximum of 3 insufflations at a time will be required. Dosing will be flexible between 8 IU/day and 80 IU/day, typically in two divided doses delivered in the morning and in the afternoon. Doses will typically increase by 8 IU twice daily (BID) at week 2 and weeks 4 and 8 until achieving the target dose of 24 IU BID at week 8. Subsequently doses may be increased in 8 IU BID increments ONLY at each visit until a maximum dose of 40 IU BID is achieved.Each bottle's label will have its own unique nonsequential randomly assigned number and not a lot number to facilitate masking. During the open label phase after approximately March 2019 the study used only the 24 IU /0.10 ml formulation and the maximum dose was 72 IU per day.
- Placebo Nasal Spray: Double-blind Phase; Placebo Nasal Spray: Open Label Phase: Placebo
  Placebo Nasal Spray: This nasal spray will contain all of the ingredients that are in the active oxytocin spray in the same quantities, except there will be no oxytocin added to the solution. It will be packaged using the same container system as the active oxytocin nasal spray. Each bottle's label will have its own unique nonsequential randomly assigned number and not a lot number to facilitate masking. Dose titration will occur using exactly the same criteria and procedures as for active study drug.
Arm/Group | Oxytocin Nasal Spray: Double-blind Phase | Placebo Nasal Spray: Double-blind Phase | Oxytocin Nasal Spray: Open Label Phase | Placebo Nasal Spray: Open Label Phase
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/144 | 1/127 | 0/122
Serious Adverse Events (participants affected / at risk) | 2/146 | 1/144 | 4/127 | 0/122
Other Adverse Events (participants affected / at risk) | 120/146 | 120/144 | 91/127 | 92/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxytocin Nasal Spray: Double-blind Phase (N=146) | Placebo Nasal Spray: Double-blind Phase (N=144) | Oxytocin Nasal Spray: Open Label Phase (N=127) | Placebo Nasal Spray: Open Label Phase (N=122)
Seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphoria (Psychiatric disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0 | 0
Appendicitis (General disorders) | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxytocin Nasal Spray: Double-blind Phase (N=146) | Placebo Nasal Spray: Double-blind Phase (N=144) | Oxytocin Nasal Spray: Open Label Phase (N=127) | Placebo Nasal Spray: Open Label Phase (N=122)
Negativism (Psychiatric disorders) | 24 | 23 | 10 | 10
Aggression Or Hostility (Psychiatric disorders) | 23 | 20 | 10 | 6
Anger Or Irritability (Psychiatric disorders) | 20 | 20 | 14 | 6
Frustration (Psychiatric disorders) | 15 | 18 | 7 | 9
Crying (Psychiatric disorders) | 13 | 17 | 10 | 10
Inappropriate Affect (Psychiatric disorders) | 13 | 13 | 5 | 4
Psychomotor Hyperactivity (Psychiatric disorders) | 11 | 10 | 3 | 7
Impulse-Control Disorder (Psychiatric disorders) | 9 | 9 | 8 | 5
Anxiety (Psychiatric disorders) | 6 | 8 | 2 | 5
Disturbance In Attention (Psychiatric disorders) | 9 | 4 | 3 | 4
Mood Swings (Psychiatric disorders) | 3 | 10 | 4 | 3
Obsessive Rumination (Psychiatric disorders) | 4 | 6 | 3 | 3
Apathy Or Boredom (Psychiatric disorders) | 4 | 5 | 5 | 4
Depressed Mood (Psychiatric disorders) | 3 | 5 | 3 | 3
Perseveration (Psychiatric disorders) | 2 | 6 | 1 | 3
Tic (Psychiatric disorders) | 3 | 4 | 5 | 4
Nightmares (Psychiatric disorders) | 3 | 3 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 2 | 2 | 1
Delusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Mania Or Hypomania (Psychiatric disorders) | 1 | 0 | 0 | 0
Pressure Of Speech (Psychiatric disorders) | 1 | 0 | 2 | 1
Agitation (Nervous system disorders) | 19 | 16 | 11 | 11
Headache (Nervous system disorders) | 11 | 22 | 6 | 8
Initial Insomnia (Nervous system disorders) | 14 | 19 | 5 | 12
Sedation (Nervous system disorders) | 19 | 12 | 5 | 8
Stereotypy (Nervous system disorders) | 13 | 8 | 3 | 5
Terminal Insomnia (Nervous system disorders) | 10 | 11 | 1 | 4
Middle Insomnia (Nervous system disorders) | 6 | 12 | 1 | 4
Restlessness (Nervous system disorders) | 11 | 3 | 4 | 3
Hypersomnia (Nervous system disorders) | 3 | 3 | 1 | 1
Confusional State (Nervous system disorders) | 1 | 2 | 2 | 0
Speech Disorder (Nervous system disorders) | 2 | 1 | 1 | 1
Dyskinesia (Nervous system disorders) | 1 | 1 | 0 | 0
Dystonia (Nervous system disorders) | 1 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Ganglion Cyst (Nervous system disorders) | 1 | 0 | 0 | 0
Photophobia (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0
Seizure Or Convulsion (Nervous system disorders) | 0 | 0 | 2 | 0
Coordination Abnormal (Nervous system disorders) | 0 | 0 | 0 | 1
Sleep Walking (Nervous system disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 53 | 67 | 33 | 33
Diarrhea (Gastrointestinal disorders) | 13 | 15 | 6 | 3
Abdominal Pain Or Discomfort (Gastrointestinal disorders) | 6 | 14 | 6 | 7
Vomiting Or Nausea (Gastrointestinal disorders) | 6 | 12 | 7 | 8
Constipation (Gastrointestinal disorders) | 7 | 9 | 4 | 6
Stomatitis (Gastrointestinal disorders) | 3 | 7 | 0 | 0
Tooth Disorder (Gastrointestinal disorders) | 3 | 5 | 3 | 3
Encopresis (Gastrointestinal disorders) | 3 | 4 | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 23 | 14 | 9 | 10
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 13 | 7 | 5
Abnormal Weight Gain (Metabolism and nutrition disorders) | 11 | 9 | 8 | 8
Abnormal Weight Loss (Metabolism and nutrition disorders) | 10 | 5 | 2 | 4
Thirst (Metabolism and nutrition disorders) | 8 | 4 | 10 | 3
Rash (Skin and subcutaneous tissue disorders) | 16 | 14 | 15 | 9
Acne (Skin and subcutaneous tissue disorders) | 5 | 12 | 4 | 6
Eczema (Skin and subcutaneous tissue disorders) | 7 | 4 | 7 | 7
Wart (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 18 | 9 | 13
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Rhinitis Nos (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Energy Increased (General disorders) | 14 | 5 | 4 | 4
Fatigue (General disorders) | 8 | 8 | 1 | 6
Pyrexia (General disorders) | 9 | 7 | 2 | 6
Swelling (General disorders) | 3 | 2 | 0 | 1
Asthenia (General disorders) | 2 | 2 | 0 | 0
Chest Pain Or Discomfort (General disorders) | 2 | 1 | 3 | 0
Night Sweats (General disorders) | 0 | 0 | 1 | 0
Allergic Hypersensitivity (Immune system disorders) | 14 | 15 | 10 | 2
Enuresis (Renal and urinary disorders) | 3 | 16 | 7 | 8
Pollakiuria (Renal and urinary disorders) | 5 | 6 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition Frequency Decreased (Renal and urinary disorders) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 8 | 6 | 13 | 7
Intentional Self-Injury (Injury, poisoning and procedural complications) | 5 | 6 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ear Ache (Ear and labyrinth disorders) | 7 | 9 | 2 | 2
Ear Congestion (Ear and labyrinth disorders) | 4 | 4 | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Epistaxis (Vascular disorders) | 11 | 10 | 6 | 4
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Libido Increased (Reproductive system and breast disorders) | 7 | 6 | 6 | 5
Breast Pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 1
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 2 | 0 | 1
Blepharospasm (Eye disorders) | 2 | 3 | 0 | 1
Dry Eye (Eye disorders) | 3 | 1 | 2 | 1
Eye Discomfort (Eye disorders) | 1 | 1 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 1 | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Growing Pains (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Specific Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Dizziness (Cardiac disorders) | 1 | 2 | 1 | 2
Cardiac Rhythm Abnormality (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 2 | 0
Enamel Discoloration (General disorders) | 0 | 1 | 0 | 0
Pituitary Analyses Anterior (Investigations) | 0 | 1 | 0 | 0
Abnormal Urinalysis (Investigations) | 0 | 0 | 1 | 0
Thrombocytopenia (Investigations) | 0 | 0 | 1 | 0
Precocious Puberty (Endocrine disorders) | 1 | 0 | 0 | 0
Skeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT01944046/Prot_SAP_001.pdf